CLINICAL TRIAL: NCT01128101
Title: Assessment of the Effects of the Combination of Spironolactone to Conventional Pharmacotherapy in Dialysis Patients
Brief Title: Effects of Spironolactone in Dialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Principal Investigator, Greicy Mara Mengue Feniman De Stefano, MSc, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-43; 3439-2010 (Other: Research Ethics Committee - Unesp)
Record Dates: First submitted 2010-05-16; First posted 2010-05-21 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Renal Failure
Keywords: spironolactone; chronic kidney disease; dialysis; LHV
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spironolactone (Experimental): The group who receive spironolactone, the dose employed will be 25 mg each other day and titrated to 25 mg daily according to potassium.
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — The group who receive spironolactone, the dose employed will be 25 mg each other day and titrated to 25 mg daily according to potassium.

SUMMARY:
Several studies indicate that chronic kidney disease patients give a high cardiovascular risk and have an intrinsic relationship with hypertension and cardiomyopathy: characterized by left ventricular hypertrophy and interstitial fibrosis. The reversal of left ventricular hypertrophy is associated with increased life expectancy in these patients. The renin angiotensin aldosterone system plays an important role in blood pressure control. Even patients using converting enzyme inhibitors inhibitors or angiotensin II blockers may experience the so called aldosterone breakthrough phenomenon (inappropriately called aldosterone escape). This phenomenon is documented in patients with heart disease and in chronic kidney disease. Spironolactone is a synthetic steroid that acts as an antagonist of aldosterone, which has historically avoided in chronic kidney disease patients, given the risk of hyperkalemia. However, its active metabolite, canrenone and spironolactone, are able to antagonize the binding of ouabain, a Na+/K+ATPase inhibitor, to its receptor. The Na+/K+-ATPase inhibition results in changes in sodium gradients, and increases the calcium influx through the transporter Na+/Ca+ in specific regions of the membrane. Spironolactone and canrenone in previous research were able to reverse left ventricular hypertrophy in chronic kidney disease patients on conservative treatment, which turn this drug and its metabolite potential tools for reversion of left ventricular hypertrophy in chronic kidney disease. The aim of this study is to verify the safety, tolerability and efficacy in the reversal of target organ damage from the use of spironolactone added to conventional antihypertensive therapy in chronic kidney disease patients on hemodialysis, in addition to measuring its ability to reduce left ventricular hypertrophy and arterial stiffness indices. Interventional randomized, double-blind, placebo-controlled study comprising two groups: one that will take 25mg of spironolactone associated with conventional antihypertensive therapy and another that will take spironolactone placebo associated with conventional antihypertensive therapy. Each group will consist of 30 patients. Clinical and laboratory investigations, as well as home monitoring of blood pressure, echocardiography, determination of pulse wave velocity, augmentation index, and central blood pressure measurement of serum aldosterone will be are evaluated before and after treatment that will last 12 months.

DETAILED DESCRIPTION:
Materials and Methods: will be conducted an interventional, randomized, double-blind, placebo-controlled study. The series will consist of patients with at least 18 years old, suffering from chronic kidney disease stage V on dialysis and mean residential blood pressure superior to 135 x 85 mm Hg with left ventricular mass indexed for height to the 2.7 power greater than 51 g/m2,7. This protocol follows the guidelines of resolution 196/96 of the Brazilian National Health Council and is approved by the Ethics Committee of the Faculty of Medicine of Botucatu - UNESP Protocol (CEP 3439-2010).

All patients will give informed consent in writing. Exclusion criteria will be thew following: history or evidence of angina or myocardial infarction, heart failure, peripheral vascular disease, Hyperkalemia, valvular disease, atrial fibrillation, anemia (hemoglobin <10 g / dl) doses of parathyroid hormone (PTH) greater than 300 pg / mL, patients in treatment with spironolactone and Patients who have suspended or initiated the use of inhibitors of angiotensin converting enzyme inhibitors, angiotensin receptor blockers and renin blockers in the last six months. Patients will be assessed at baseline (before the run-in phase), weekly in the first month and monthly thereafter until one year, or 52 weeks. Will be include clinical examination at each visit and laboratory tests. In the visits of weeks zero, 26 and 52 will be held monitoring home blood pressure, echocardiography, determining the of pulse wave velocity, central arterial pressure and augmentation index. Aldosterone an ouabaín will be monitored immediately before run-in fase and at 52 weeks.

Groups: Patients will be randomly divided into two groups: active drug and placebo groups. One group will receive spironolactone and the other placebo spironolactone. It is important to note that placebo therapy is only of spironolactone and not other anti-hypertensive drugs, so patients will not in any way deprived of the benefit established in the literature which is the reduction of blood pressure. Physicians' assistants enrolled will be free to prescribe any antihypertensive medication except the study drug. In the active treatment group, the dose employed will be 25 mg each other day and titrated to 25 mg daily according to the potassium. Patients with potassium between 5.5 and 5.9 mmol/L will have reduced spironolactone to 25 mg each other day if they are in use 25 mg daily or will not increase the dose. These patients receive pharmaceutical care and nutritional guidance according the routine of the unit.

The placebo group will receive placebo with the same protocol. These patients also receive pharmaceutical care and nutritional guidance, beyond any conventional antihypertensive treatment. The pharmaceutical form of placebo will consist of colloidal silicon dioxide, cornstarch, lactose monohydrate, microcrystalline cellulose and magnesium stearate, inert excipients according to reference literature. The pharmaceutical form of the active drug will consist of spironolactone 25 mg and the other components of the placebo.

The laboratory tests will be performed as routine in our dialysis unit, which follow the rules of operation of hemodialysis established by the Brazilian Ministry of Health, as follows: blood samples are collected immediately before the start of hemodialysis for routine hematology (red blood cells, platelets white blood cell count) and biochemical (urea, creatinine, potassium, calcium, phosphorus, glutamic-pyruvic transaminase and venous blood gas) monthly. Will be held quarterly glycosylated hemoglobin for diabetics, total proteins and fractions, alkaline phosphatase, transferrin, serum iron, ferritin, C-reactive protein, parathyroid hormone and lipid levels, the dosage of uric acid is each six months and aluminum will be annual. Measurement of plasma renin, aldosterone, angiotensin II and ouabaín will be held at time zero and after 52 weeks. Urine collections in 24 hours will be obtained for measurement of residual urea clearance and calculation of protein nitrogen appearance in weeks zero, 26 and 52. Will be collected monthly samples of urine after dialysis for determination of fractional clearance of urea (dialysis dose) that will be determined by the Daugirdas's formula (1995). Prior to collecting samples for measurement of plasma renin, the patient should be 2 h in the supine position (stabilization of serum and standardization of interpretation of results).

Blood samples for determination of potassium will be collected weekly in the first four weeks, fortnightly during the second month and thereafter will be held monthly dosages. All antihypertensive medications will be maintained and titrated according to patients' needs to achieve the target of 135x85 mm Hg in residential blood pressure monitoring. Criteria for suspension therapy: patients are withdrawn from the protocol if develop severe hyperkalemia, defined as one serum potassium concentration equal or superior than 6.5 mmol/L in an isolated or repeated measures equal to or greater than 6.0 mmol/L. Each death will be analyzed by an independent committee and in the event of a statistical difference in the mortality of active drug compared to placebo, the work will be suspended immediately.

Echocardiography: The procedure for echocardiography will be performed according to previously standardized technique. The following data are recorded: heart rate, systolic and diastolic pressures obtained during the examination, systolic and diastolic dimensions of left ventricular posterior wall thickness and septum, internal dimensions of left atrium and aorta, stroke volume, ejection time of LV peak mitral flow velocity (E), peak velocity of atrial filling (A), deceleration time of E wave; slope of the deceleration ramp of the E wave and isovolumic relaxation time. These data will be used to calculate the relative thickness of the left ventricle, the left atrium/aortic diameter, left ventricular mass index, left ventricular mass, fractional shortening of the ventricular diameter, meridian end-systolic stress, cardiac output index, heart rate, left ventricular stroke work.

Home monitoring of blood pressure: will be conducted with equipment validated by the BHS and AAMI (Omron model HEM 781 INT). Patients will receive guidance to carry out three measurements in the morning upon waking and fasting and three measures at bedtime during a week exempting Saturday and Sunday. The measures will be undertaken with the patient seated, back supported, arm at heart level, the forearm in the supine position. Will use the upper limb that showed the highest blood pressure measurement in the office, except if the patient has vascular access in one of the arms which will require taking the measurements in the contralateral arm. The patient will be instructed to not perform measurements of any other person with the same apparatus. After one week the patient will bring the unit back and the device memory will be analyzed. Will be taken as representative value of the average home blood pressure of all valid measurements, except for the first day.

Pulse wave velocity, central arterial blood pressure and augmentation index will be performed by applanation tonometry. The patient should be fasting on exam day and will remain at rest for five minutes before the start. The analysis of PWV will be held simultaneously with checking blood pressure. Begins the reading with the placement of the forearm without arteriovenous fistula on support equipment, palpation to the radial artery and apply the tonometer sensor. The corresponding central waveform is generated by the use of a validated transfer function (SphygmoCor, AtCor Medical, Sydney, Australia). Will be collected waves pulse for 10 seconds at least twice, which will be recorded directly on a laptop. After at least 20 recorded waveforms, the average of peripheral, as well as their corresponding central, and also an average of measurements of systolic, diastolic and pulse pressure.

Statistical analysis: The sample size of 24 patients in each group (active drug and placebo groups) is sufficient to detect a difference of 15g/m2 in left ventricular mass index with standard deviation of the differences estimated in 23g/m2, statistical power of 0.8 and p <0.05. However, as the expected mortality of up to 20% per year, the total sample is comprised of 30 patients in each group. The results will be quantified and analyzed descriptively, initially through the observation of minimum and maximum values, and the calculation of averages and their standard deviations. To investigate the behavior of groups, will be used the techniques of analysis of variance parametric and nonparametric, followed by a posteriorly tests appropriate to the characteristics of each variable evaluated.

ELIGIBILITY:
Inclusion Criteria:

The series will consist of:

1. Patients with at least 18 years of age,
2. Suffering from chronic kidney disease stage V on dialysis,
3. Mean blood pressure residential than 135 x 85 mm Hg and
4. Who present left ventricular mass indexed for height to the 2.7 power greater than 51 g/m2, 7.

Exclusion Criteria:

1. History or evidence of angina or myocardial infarction,
2. Heart failure,
3. Peripheral vascular disease,
4. Hyperkalemia
5. Previous valve atrial fibrillation,
6. Anemia (hemoglobin <10 g/dl),
7. Doses of parathyroid hormone (PTH) greater than 300 pg/mL,
8. Patients being treated with spironolactone and
9. Patients who have suspended or initiated the use of inhibitors of angiotensin converting enzyme inhibitors, angiotensin receptor blockers (ARBs) renin blockers in the last six months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of Left Ventricular Hypertrophy | 12 months
  The reduction of left ventricular hypertrophy will be measured by echocardiography, blood pressure monitoring residential and pulse wave velocity.

SECONDARY OUTCOMES:
To evaluate the safety and efficacy of the use of spironolactone at a dose of 25mg in patients with chronic kidney disease on hemodialysis. | 12 months
  Measurement of serum potassium and other routine laboratory parameters pertaining to the hemodialysis unit of the Hospital of the Medical School of Botucatu - UNESP.

CONTACTS AND LOCATIONS:
Overall Officials: Luis C Martin, Doctor, Study Director — UPECLIN HC FM Botucatu Unesp
Locations (1):
- Hospital of the Medical School of Botucatu, Botucatu, São Paulo, Brazil

REFERENCES:
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138
- [Derived] Feniman De Stefano GM, Zanati-Basan SG, De Stefano LM, Silva VR, Xavier PS, Barretti P, da Silva Franco RJ, Caramori JC, Martin LC. Aldosterone is associated with left ventricular hypertrophy in hemodialysis patients. Ther Adv Cardiovasc Dis. 2016 Oct;10(5):304-13. doi: 10.1177/1753944716644583. Epub 2016 Apr 27. PMID 27122492
- [Derived] Feniman-De-Stefano GM, Zanati-Basan SG, De Stefano LM, Xavier PS, Castro AD, Caramori JC, Barretti P, Franco RJ, Martin LC. Spironolactone is secure and reduces left ventricular hypertrophy in hemodialysis patients. Ther Adv Cardiovasc Dis. 2015 Aug;9(4):158-67. doi: 10.1177/1753944715591448. Epub 2015 Jun 26. PMID 26116627